CLINICAL TRIAL: NCT02130622
Title: A Pilot, Randomized, Double-blind, Placebo-controlled Trial of Promethazine for Treatment of Diabetic Gastroparesis.
Brief Title: Study of Promethazine for Treatment of Diabetic Gastroparesis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D14076
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Gastroparesis
Keywords: Diabetic Gastroparesis; Promethazine
MeSH Terms: interventions — Promethazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Promethazine (Experimental): Promethazine 12.5 mg P.O. t.i.d. for 4 weeks
  Interventions: Drug: Promethazine
- Sugar Pill (Placebo Comparator): Placebo P.O. t.i.d. for 4 weeks
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Promethazine
  Other Names: Phenergan
  Arms: Promethazine
Drug: Sugar pill
  Other Names: Placebo
  Arms: Sugar Pill

SUMMARY:
Adult diabetic patients (ages 18-65) with gastric emptying scintigraphy-confirmed delayed gastric emptying will be recruited to participate in the study. Using double-blinded methodology, study participants will be randomly assigned to one of two treatment arms: promethazine 12.5 mg three times daily for 28 days or placebo three times daily for 28 days. The primary outcome will be the change in gastroparesis symptom severity, as measured by the Gastroparesis Cardinal Symptom Index (GCSI) at four weeks compared to baseline. Participants will be seen for a clinic evaluation at weeks 0, 2 and 4, during which symptom scores, adverse events and treatment compliance will be assessed. It is hypothesized promethazine treatment will be superior to placebo in improving symptoms of gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-65 years of age
* clinical diagnosis of diabetic gastroparesis.
* EGD without evidence of gastric outlet obstruction within the past five years
* gastric emptying scintigraphy test demonstrating >10% solid food retention at 4 hours within the past three years.

Exclusion Criteria:

* the inability or unwillingness to provide informed consent
* currently pregnant or breast feeding
* prior placement of a gastric stimulator
* pyloric botulinum toxin injection within the past 12 months
* prior gastric surgery
* history of a connective tissue disorder
* use of narcotic medication within the past four weeks
* hemoglobin A1C >12 mg/dL within the past 3 months
* current or recent (within past 4 weeks) use of promethazine, metoclopramide or domperidone
* hypersensitivity or prior adverse reaction to promethazine
* concomitant use of phenothiazines (i.e. prochlorperazine, chlorpromazine) or other agents likely to increase extrapyramidal reactions
* concomitant use of tiotropium or ipratropium
* narrow angle glaucoma
* urinary retention
* Parkinson's disease
* significant psychiatric disease
* history of seizure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian E. Lacy, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Cherian D, Parkman HP. Nausea and vomiting in diabetic and idiopathic gastroparesis. Neurogastroenterol Motil. 2012 Mar;24(3):217-22, e103. doi: 10.1111/j.1365-2982.2011.01828.x. Epub 2011 Nov 27. PMID 22118574
- [Background] Janssen P, Harris MS, Jones M, Masaoka T, Farre R, Tornblom H, Van Oudenhove L, Simren M, Tack J. The relation between symptom improvement and gastric emptying in the treatment of diabetic and idiopathic gastroparesis. Am J Gastroenterol. 2013 Sep;108(9):1382-91. doi: 10.1038/ajg.2013.118. PMID 24005344
- [Background] Ricci DA, Saltzman MB, Meyer C, Callachan C, McCallum RW. Effect of metoclopramide in diabetic gastroparesis. J Clin Gastroenterol. 1985 Feb;7(1):25-32. doi: 10.1097/00004836-198502000-00003. PMID 3884697
- [Background] McCallum RW, Ricci DA, Rakatansky H, Behar J, Rhodes JB, Salen G, Deren J, Ippoliti A, Olsen HW, Falchuk K, et al. A multicenter placebo-controlled clinical trial of oral metoclopramide in diabetic gastroparesis. Diabetes Care. 1983 Sep-Oct;6(5):463-7. doi: 10.2337/diacare.6.5.463. PMID 6400707
- [Background] Perkel MS, Moore C, Hersh T, Davidson ED. Metoclopramide therapy in patients with delayed gastric emptying: a randomized, double-blind study. Dig Dis Sci. 1979 Sep;24(9):662-6. doi: 10.1007/BF01314461. PMID 385260
- [Background] Snape WJ Jr, Battle WM, Schwartz SS, Braunstein SN, Goldstein HA, Alavi A. Metoclopramide to treat gastroparesis due to diabetes mellitus: a double-blind, controlled trial. Ann Intern Med. 1982 Apr;96(4):444-6. doi: 10.7326/0003-4819-96-4-444. PMID 7065559
- [Background] Patterson D, Abell T, Rothstein R, Koch K, Barnett J. A double-blind multicenter comparison of domperidone and metoclopramide in the treatment of diabetic patients with symptoms of gastroparesis. Am J Gastroenterol. 1999 May;94(5):1230-4. doi: 10.1111/j.1572-0241.1999.00456.x. PMID 10235199
- [Background] Erbas T, Varoglu E, Erbas B, Tastekin G, Akalin S. Comparison of metoclopramide and erythromycin in the treatment of diabetic gastroparesis. Diabetes Care. 1993 Nov;16(11):1511-4. doi: 10.2337/diacare.16.11.1511. PMID 8299441
- [Background] McHugh S, Lico S, Diamant NE. Cisapride vs metoclopramide. An acute study in diabetic gastroparesis. Dig Dis Sci. 1992 Jul;37(7):997-1001. doi: 10.1007/BF01300277. PMID 1618070
- [Background] Feldman M, Smith HJ. Effect of cisapride on gastric emptying of indigestible solids in patients with gastroparesis diabeticorum. A comparison with metoclopramide and placebo. Gastroenterology. 1987 Jan;92(1):171-4. doi: 10.1016/0016-5085(87)90854-7. PMID 3781184
- [Background] Ehrenpreis ED, Deepak P, Sifuentes H, Devi R, Du H, Leikin JB. The metoclopramide black box warning for tardive dyskinesia: effect on clinical practice, adverse event reporting, and prescription drug lawsuits. Am J Gastroenterol. 2013 Jun;108(6):866-72. doi: 10.1038/ajg.2012.300. PMID 23735907
- [Background] Tan PC, Khine PP, Vallikkannu N, Omar SZ. Promethazine compared with metoclopramide for hyperemesis gravidarum: a randomized controlled trial. Obstet Gynecol. 2010 May;115(5):975-981. doi: 10.1097/AOG.0b013e3181d99290. PMID 20410771
- [Background] Braude D, Crandall C. Ondansetron versus promethazine to treat acute undifferentiated nausea in the emergency department: a randomized, double-blind, noninferiority trial. Acad Emerg Med. 2008 Mar;15(3):209-15. doi: 10.1111/j.1553-2712.2008.00060.x. PMID 18304050
- [Background] Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Development and validation of a patient-assessed gastroparesis symptom severity measure: the Gastroparesis Cardinal Symptom Index. Aliment Pharmacol Ther. 2003 Jul 1;18(1):141-50. doi: 10.1046/j.1365-2036.2003.01612.x. PMID 12848636
- [Background] Revicki DA, Camilleri M, Kuo B, Szarka LA, McCormack J, Parkman HP. Evaluating symptom outcomes in gastroparesis clinical trials: validity and responsiveness of the Gastroparesis Cardinal Symptom Index-Daily Diary (GCSI-DD). Neurogastroenterol Motil. 2012 May;24(5):456-63, e215-6. doi: 10.1111/j.1365-2982.2012.01879.x. Epub 2012 Jan 27. PMID 22284754
- [Background] Reilly MC, Bracco A, Ricci JF, Santoro J, Stevens T. The validity and accuracy of the Work Productivity and Activity Impairment questionnaire--irritable bowel syndrome version (WPAI:IBS). Aliment Pharmacol Ther. 2004 Aug 15;20(4):459-67. doi: 10.1111/j.1365-2036.2004.02091.x. PMID 15298641
- [Background] Wahlqvist P, Carlsson J, Stalhammar NO, Wiklund I. Validity of a Work Productivity and Activity Impairment questionnaire for patients with symptoms of gastro-esophageal reflux disease (WPAI-GERD)--results from a cross-sectional study. Value Health. 2002 Mar-Apr;5(2):106-13. doi: 10.1046/j.1524-4733.2002.52101.x. PMID 11918826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the gastroenterology clinic at Dartmouth-Hitchcock Medical Center at the time of routine appointments.
Groups:
- Promethazine: Promethazine 12.5 mg P.O. t.i.d. for 4 weeks
  Promethazine
- Sugar Pill: Placebo P.O. t.i.d. for 4 weeks
  Sugar pill
Period: Overall Study
Arm/Group | Promethazine | Sugar Pill
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Promethazine | Sugar Pill | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-reported Symptoms as Measured by the Gastroparesis Cardinal Symptom Index Score (GCSI, 14) From Week 0 to Week 4.
Time Frame: 4 weeks
Population: Insufficient recruitment resulting in insufficient data to analyze
Arm/Group | Promethazine | Sugar Pill
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Occurrence of Adverse Events
Time Frame: 4 weeks
Population: Insufficient recruitment resulting in insufficient data to analyze
Arm/Group | Promethazine | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Use of Rescue Medication
Description: Frequency of use of the "rescue medication" meclizine
Time Frame: 4 weeks
Population: Data not collected
Arm/Group | Promethazine | Sugar Pill
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The Impact on Work Activity as Measured by the Work Productivity and Activity Impairment Questionnaire. (WPAI).
Time Frame: 4 weeks
Population: Insufficient recruitment resulting in insufficient data to analyze
Arm/Group | Promethazine | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of ICF signature through study completion, approximately 5 weeks
Arm/Group | Promethazine | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Promethazine (N=2) | Sugar Pill (N=1)
Auditory Hallucinations (Psychiatric disorders) | 1 (2) | 0 (0)
Nightmares (Psychiatric disorders) | 1 (3) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Insufficient enrollment to provide study results. Study terminated before full enrollment due to lack of participant interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No